CLINICAL TRIAL: NCT02893592
Title: Efficiency, Predictability and Security of the Trans-epithelial Photorefractive Keratectomy (Trans-PRK) for Low and Medium Myopia and Astigmatism: Retrospective Study About 118 Eyes
Brief Title: Efficiency, Predictability and Security of the Trans-epithelial Photorefractive Keratectomy
Acronym: MYOPAS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-11Obs-CHRMT
Record Dates: First submitted 2016-08-30; First posted 2016-09-08 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-08

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The photorefractive keratectomy was the first correction mode refractive laser. It's a photo-ablation of a predetermined thickness of anterior corneal stroma. Debridement of epithelium can be done either mechanically (m-PRK) or by laser (trans-PRK). Trans-PRK has a lot of interests: facility and speed of procedure as well as suppression of human variable. Very good results are obtained by m-PRK. The aim of this study is to show equivalence or non inferiority of trans-PRK over conventional m-PRK in terms of safety and refractive efficiency

ELIGIBILITY:
Inclusion Criteria:

* patients with stable refractive error (more than 2 years)
* Myopia up to -4.00 diopters and astigmatism up to -3.00 diopters

Exclusion Criteria:

* Phototherapeutic keratectomy (PTK)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Were included patients with myopia up to -4D (dioptries) and cylinders up to -3D.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2015-10; Primary Completion 2015-11 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
visual acuity | Month 2
  LogMar

IPD SHARING:
Plan to Share IPD: No